CLINICAL TRIAL: NCT06537310
Title: An Open-label, Multicenter, Dose-escalation, Randomized, Phase I Study to Evaluate Safety, Pharmacokinetics, Pharmacodynamics and Anti-Tumor Activity of RO7567132, as a Single Agent and in Combination With Atezolizumab in Participants With Advanced and/or Metastatic Solid Tumors
Brief Title: A Dose-escalation Study of RO7567132 as Single Agent and in Combination With Atezolizumab in Participants With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BP44956; 2024-512839-70-00 (Other: EU Trial Number)
Record Dates: First submitted 2024-08-01; First posted 2024-08-05 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Cancer-Neoplasms
MeSH Terms: interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part I: RO7567132 Dose Escalation With or Without Atezolizumab (Experimental)
  Interventions: Drug: RO7567132 and Atezolizumab
- Part II: RO7567132 Backfill With Atezolizumab (Experimental)
  Interventions: Drug: RO7567132 and Atezolizumab

INTERVENTIONS:
Drug: RO7567132 and Atezolizumab — RO7567132 will be administered either as monotherapy or in combination with atezolizumab at a dose and schedule as specified for the respective cohort.
  Arms: Part I: RO7567132 Dose Escalation With or Without Atezolizumab
Drug: RO7567132 and Atezolizumab — RO7567132 will be administered in combination with atezolizumab at a dose and schedule as specified for the respective cohort.
  Arms: Part II: RO7567132 Backfill With Atezolizumab

SUMMARY:
The purpose of this study is to evaluate the safety, pharmacokinetics (PK), pharmacodynamics (PD) and preliminary clinical activity of RO7567132 as single agent and in combination with atezolizumab. The study will enroll adult participants with selected locally advanced and/or metastatic solid tumors for whom standard therapy does not exist, or has proven to be ineffective or intolerable.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged ≥18 years
* Body weight > 40 kilograms (kg)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 and Life expectancy of at least 12 weeks
* Participants with advanced and/or metastatic solid tumors
* Availability and willingness to provide a mandatory archival tumor specimen or (if not available) a fresh baseline biopsy
* Negative serum pregnancy test
* Participants must have adequate cardiovascular, hematological, liver and renal function.

Exclusion Criteria:

* Known central nervous system (CNS) tumors or metastases and leptomeningeal metastases
* Active second malignancy within 2 years prior to screening
* History or current clinically significant cardiovascular/cerebrovascular disease
* Active or history of autoimmune disease
* Serious, uncontrolled infection
* Known clinically significant liver disease
* Unresolved acute toxicity > grade 1 from prior therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2024-09-16 (Actual); Primary Completion 2029-06-19 (Estimated); Study Completion 2029-06-19 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) Graded According to Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE v5.0) | Up to a maximum of 27 months
Percentage of Participants With Dose-limiting Toxicities (DLTs) | From baseline to 3 weeks on study

SECONDARY OUTCOMES:
Maximum Concentration (Cmax) Derived for RO7567132 | Up to a maximum of 24 months
Time of Maximum Concentration (Tmax) | Up to a maximum of 24 months
Minimum Concentration (Cmin) | Up to maximum of 24 Months
Clearance (CL) or Apparent Clearance (CL/F) | Up to a maximum of 24 months
Volume of Distribution at Steady State (Vss) | Up to a maximum of 24 months
Area Under the Curve (AUC) for Various Time Intervals | Up to a maximum of 24 months
Percentage of Participants with Anti-Drug Antibodies (ADAs) to RO7567132 | Up to 24 months
Objective Response Rate (ORR) | Up to a maximum of 24 months
Disease Control Rate (DCR) | Up to a maximum of 24 months
Duration of Response (DoR) | Up to a maximum of 24 months
Progression Free Survival (PFS) | Up to a maximum of 24 months
Overall Survival (OS) | Up to a maximum of 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical trails, Study Director — Hoffmann-La Roche
Locations (11):
- Australia (2):
  - Kinghorn Cancer Centre, Darlinghurst, New South Wales
  - Austin Health, Heidelberg, Victoria
- UZ Leuven Gasthuisberg, Leuven, Belgium
- Canada (3):
  - BC Cancer ? Vancouver, Vancouver, British Columbia
  - Princess Margaret Cancer Center, Toronto, Ontario
  - McGill University Health Center, Montreal, Quebec
- Rigshospitalet, København Ø, Denmark
- Spain (4):
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Vall d?Hebron Institute of Oncology (VHIO), Barcelona, Barcelona
  - Clinica Universidad de Navarra Madrid, Madrid
  - Fundacion Jimenez Diaz, Madrid

IPD SHARING:
Plan to Share IPD: No